CLINICAL TRIAL: NCT00635336
Title: Phase I Study of Vaccination With MPHOSHP1 and DEPDC1 Derived Epitope Peptides for HLA-A-24-positive Patients With Advanced Bladder Cancer
Brief Title: Novel Peptide Vaccination for Patients With Advanced Bladder Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Iwate Medical University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Department of Urology, Iwate Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMU-H18-59-P1
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2009-01

CONDITIONS: Bladder Cancer
Keywords: Epitope peptide; CTL; Advanced bladder cancer; Vaccination; advanced bladder cancer which showed resistance for standard treatments
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — KIF20B protein, human; DEPDC1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: MPHOSPH1 and DEPDC1 — DEPDC1-9-294, and/or MPHOSPH1-9-278 will be administered by subcutaneously injection once every week for 3 months thereafter once two weeks. These peptides are determined to administer in accordance with the protein expression using immunohistochemical staining. These peptides are conjugated with Montanide ISA 51 as an adjuvant.

SUMMARY:
The purpose of this study is to evaluate the safety and clinical efficacy of novel vaccination for advanced bladder cancer.

DETAILED DESCRIPTION:
DEP domain containing 1(DEPDC1) and M phase phosphoprotein 1(MPHOSPH1) have been identified using genome-wide expression profile analysis by the use of cDNA microarray in our previous studies. We have determined the HLA-A*2402 restricted epitope peptides derived from DEPDC1, DEPDC1-9-294, and MPHOSPH1, MPHOSPH1-9-278. These epitopes showed strong IFN-g production when stimulated with the appropriate targets expressed the appropriate protein and HLA-A*2402. Furthermore, when vaccinated these peptides, specific CTLs were determined after the vaccination. Therefore we focused on the safety and efficacy of novel vaccination for the advanced bladder cancer patients who already showed resistance to standard chemotherapies or radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS

1. advanced bladder cancer which already showed resistance to standard treatments
2. Protein expression of MPHOSPH1 and DEPDC1 on the tumor

PATIENTS CHARACTERISTICS

1. Patients who showed resistance to standard chemotherapies or radiotherapy
2. Histological diagnosis is transitional cell carcinoma
3. HLA-A*2402
4. ECOG performance status of 0 to 1
5. Age ≥ 20 years, ≤80 years
6. WBC≥ 2,000/mm³, ≤15000/mm³ Platelet count ≥ 75000/mm³ AST, ALT ≤150 IU/l Total bilirubin ≤ 3.0 mg/dl Creatinine ≤ 3.0 mg/dl
7. lesion of bladder cancer must express MPHOSPH1 or DEPDC1
8. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
2. Breastfeeding
3. Patients willing to childbearing ( Refusal or inability to use effective means of contraception)
4. Serious infections requiring antibiotics
5. Concomitant treatment with steroids or immunosuppressing agent
6. Other malignancy difficult to control.
7. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-02; Primary Completion 2007-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
feasibility (toxicities as assessed by NCI-CTCAE version 3) | 3 years

SECONDARY OUTCOMES:
objective response rate as assessed by RECIST criteria | 3 years
CTL response | 3 years
CD8 population | 3 years
Change in level of regulatory T cells | 3 years
survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tomoaki Fujioka, M.D. & Ph.D., Study Chair — Department of Urology, Iwate Medical University
Locations (1):
- Iwate Medical University School of Medicine, Morioka, Iwate, Japan

REFERENCES:
- [Background] Rosenberg SA, Lotze MT, Yang JC, Aebersold PM, Linehan WM, Seipp CA, White DE. Experience with the use of high-dose interleukin-2 in the treatment of 652 cancer patients. Ann Surg. 1989 Oct;210(4):474-84; discussion 484-5. doi: 10.1097/00000658-198910000-00008. PMID 2679456
- [Background] Okabe H, Satoh S, Kato T, Kitahara O, Yanagawa R, Yamaoka Y, Tsunoda T, Furukawa Y, Nakamura Y. Genome-wide analysis of gene expression in human hepatocellular carcinomas using cDNA microarray: identification of genes involved in viral carcinogenesis and tumor progression. Cancer Res. 2001 Mar 1;61(5):2129-37. PMID 11280777
- [Background] Hasegawa S, Furukawa Y, Li M, Satoh S, Kato T, Watanabe T, Katagiri T, Tsunoda T, Yamaoka Y, Nakamura Y. Genome-wide analysis of gene expression in intestinal-type gastric cancers using a complementary DNA microarray representing 23,040 genes. Cancer Res. 2002 Dec 1;62(23):7012-7. PMID 12460921
- [Background] Bienz M, Clevers H. Linking colorectal cancer to Wnt signaling. Cell. 2000 Oct 13;103(2):311-20. doi: 10.1016/s0092-8674(00)00122-7. No abstract available. PMID 11057903
- [Result] Kanehira M, Katagiri T, Shimo A, Takata R, Shuin T, Miki T, Fujioka T, Nakamura Y. Oncogenic role of MPHOSPH1, a cancer-testis antigen specific to human bladder cancer. Cancer Res. 2007 Apr 1;67(7):3276-85. doi: 10.1158/0008-5472.CAN-06-3748. PMID 17409436
- [Result] Kanehira M, Harada Y, Takata R, Shuin T, Miki T, Fujioka T, Nakamura Y, Katagiri T. Involvement of upregulation of DEPDC1 (DEP domain containing 1) in bladder carcinogenesis. Oncogene. 2007 Sep 27;26(44):6448-55. doi: 10.1038/sj.onc.1210466. Epub 2007 Apr 23. PMID 17452976